CLINICAL TRIAL: NCT01488825
Title: Effect of Yoga Intervention on Episodic Tension Type Headache: A Randomized Controlled Trial
Brief Title: Yoga Intervention Study on Episodic Tension Type Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMP-0090-YR
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Episodic Tension Type Headache
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait-list control group (No Intervention): The wait-list control group received no intervention, or instruction and they were observed with their usual care for 12-weeks intervention period. Upon completion of the study, this group received 12 weeks of yoga intervention.
- Yoga Intervention Group (Experimental): The yoga sessions developed specifically for study participant consisted of 12 weekly 60-minute designed to benefit in episodic tension type headache.
  Interventions: Behavioral: Yoga Therapy

INTERVENTIONS:
Behavioral: Yoga Therapy — Therapeutically oriented style of yoga originated from Pancha Kosha philosophy of Vedanta was used throughout the trial. All the sessions emphasized on postures, breathing practices with the specific focus on relaxation, combination of chants and meditation. Once a week, Kunjal and Jalaneti (cleansing practices) were practiced in guidance of therapist. They all were instructed to eat light and rest on Kriya days.
  Arms: Yoga Intervention Group

SUMMARY:
The present study was designed to evaluate effect of yoga intervention on patients having frequent tension type headache.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 to 60 years
* more than 5 but fewer than 15 headache episodes per month
* headache intensity moderate to severe

Exclusion Criteria:

* Patients on anti-psychotic, antidepressant or any prophylactic medication
* pregnancy
* Taking psychotherapy or any other alternative medicine
* migraine headache more than 1 day a month
* pain disorder, psychiatric or medical disorder requiring immediate treatment,
* headache due to sinusitis, eyestrain, cervical spondylosis and posttraumatic headaches

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2005-01; Primary Completion 2006-02 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Frequency of headache | 3 Months

SECONDARY OUTCOMES:
Duration of Headache | 3 months
Severity of headache | 3 Months
Analgesic consumption | 3 Months
Anxiety levels | 3 months
Depression | 3 months
Stress | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Neha SHARMA, PhD, Principal Investigator — NMP Medical Research Institute
Locations (1):
- Pain Clinic, NMP Medical Research Institute, Jaipur, Rajasthan, India